CLINICAL TRIAL: NCT03215342
Title: Cognitive Rehabilitation in Pediatric Acquired Brain Injury - a Randomized Controlled Trial
Brief Title: Cognitive Rehabilitation in Pediatric Acquired Brain Injury
Acronym: CORE-pABI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/772
Record Dates: First submitted 2017-07-11; First posted 2017-07-12 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Brain Injuries
Keywords: Child; Rehabilitation; Psychotherapy, groups
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pGMT (Experimental): Pediatric Goal Management Training
  Interventions: Behavioral: Pediatric Goal Management Training
- pBHW (Experimental): Pediatric Brain Health Workshop
  Interventions: Behavioral: Pediatric Brain Health Workshop

INTERVENTIONS:
Behavioral: Pediatric Goal Management Training — 7 GMT modules will be administered in 7x2 hours sessions (ten groups). Manualized intervention; metacognitive strategies for improving attention and problem solving. Homework assignments between sessions.
  Other Names: GMT
  Arms: pGMT
Behavioral: Pediatric Brain Health Workshop — 7 pBHW modules will be administered in 7x2 hours sessions (ten groups). Psychoeducation; brain (dys)function, plasticity, memory, executive function, and attention. Stress, physical exercise, sleep, nutrition, and energy management. Homework assignments between sessions
  Other Names: active control condition; pBHW
  Arms: pBHW

SUMMARY:
Acquired brain injury (e.g., traumatic brain injury, brain tumour, brain infections) is one of the leading causes of death and disability for children and adolescents. Importantly, injuries affecting the brain in childhood or adolescence appear during a time of development when the brain is particularly vulnerable. Thus, pediatric acquired brain injury does not only impact cognitive functions at the time of injury or onset of disease, but also cognitive functions that are yet to develop. Changes in cognitive function, and in particular executive dysfunction due to acquired brain injury, cause significant real-life disability, yet solid evidence in support of executive functioning interventions for children and adolescents is lacking. In the present study different group-based cognitive rehabilitation interventions will be compared. The aim of the study is to investigate if a group-based "brain training" intervention is able to improve executive function in children and adolescents after acquired brain injury. Efficacy will be assessed immediately after intervention, but also six months after the intervention. The project is in line with international research efforts aimed at establishing more knowledge about how children and adolescents with brain injuries respond to cognitive rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with traumatic brain injury, brain tumor or damage by inflammation in the brain
* more than 12 months since injury/illness or more than 12 months since ended cancer therapy
* evidence of executive dysfunction in everyday life

Exclusion Criteria:

* cognitive, sensory, physical, or language impairment affecting the capacity to attend mainstream school and/or complete the training program
* pre-injury neurological disease or psychiatric disorder
* recently detected brain tumor relapse
* unfit for evaluation of outcome (independent evaluation by 2 investigators)
* not fluent in Norwegian language

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
executive function in daily life | change from baseline up to 6 months
  Behavior Rating Inventory of Executive Function (BRIEF; self, teacher and parent form

SECONDARY OUTCOMES:
Performance on Conners Continuous Performance Test III | change from baseline up to 6 months
Performance on BADS-C | change from baseline up to 6 months
Performance on D-KEFS Trail Making Test 1-4 | change from baseline up to 6 months
performance on D-KEFS Color Word Interference Test | change from baseline up to 6 months
Performance on Children's Cooking Task test | change from baseline up to 6 months
Performance on NEPSY-II Social Perception test | change from baseline up to 6 months
Score on Health Behaviour Inventory | change from baseline up to 6 months
  questionnaire
Score on Glasgow Outcome Scale Extended Pediatric | change from baseline up to 6 months
  questionnaire
Score an EQ-5D-Y | change from baseline up to 6 months
  questionnaire
Score on Family Functioning Scale | change from baseline up to 6 months
  questionnaire
Score on Center for Epidemiologic Studies Depression Scale | change from baseline up to 6 months
  questionnaire
Score on Pediatric Quality of Life Inventory | change from baseline up to 6 months
  questionnaire
Score on Cognitive Failures Questionnaire | change from baseline up to 6 months
Score on ADHD Rating Scale IV | change from baseline up to 6 months
  questionnaire
Score on Child Behavior Checklist | change from baseline up to 6 months
  questionnaire
Score on Harter Self Perception Profile for Children | change from baseline up to 6 months
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kari Risnes, md phd, Study Director — St. Olavs Hospital
Locations (2):
- Norway (2):
  - Oslo universitetssykehus HF, Oslo
  - Barne og ungdomsklinikken St Olavs Hospital, Trondheim

REFERENCES:
- [Background] Hypher RE, Brandt AE, Risnes K, Ro TB, Skovlund E, Andersson S, Finnanger TG, Stubberud J. Paediatric goal management training in patients with acquired brain injury: study protocol for a randomised controlled trial. BMJ Open. 2019 Aug 1;9(8):e029273. doi: 10.1136/bmjopen-2019-029273. PMID 31375619
- [Result] Brandt AE, Finnanger TG, Hypher RE, Ro TB, Skovlund E, Andersson S, Risnes K, Stubberud J. Rehabilitation of executive function in chronic paediatric brain injury: a randomized controlled trial. BMC Med. 2021 Nov 2;19(1):253. doi: 10.1186/s12916-021-02129-8. PMID 34724955
- [Derived] Hypher R, Brandt AE, Skovlund E, Skarbo AB, Barder HE, Andersson S, Ro TB, Risnes K, Finnanger TG, Stubberud J. Metacognitive strategy training versus psychoeducation for improving fatigue in children and adolescents with acquired brain injuries: A randomized controlled trial. Neuropsychology. 2022 Oct;36(7):579-596. doi: 10.1037/neu0000845. Epub 2022 Aug 4. PMID 35925734
- [Derived] Hypher R, Andersson S, Finnanger TG, Brandt AE, Hoorelbeke K, Lie HC, Barder HE, Larsen SM, Risnes K, Ro TB, Stubberud J. Fatigue following pediatric acquired brain injury: Interplay with associated factors in a clinical trial population compared to healthy controls. Neuropsychology. 2021 Sep;35(6):609-621. doi: 10.1037/neu0000753. Epub 2021 Jul 1. PMID 34197132

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT03215342/SAP_000.pdf